CLINICAL TRIAL: NCT02931058
Title: Efficacy of Pre-operative Quadriceps Strength Training on Knee-extension Strength Before and Shortly Following Total Knee Arthroplasty: A Randomized Dose-response Trial (The QUADX-1 Trial)
Brief Title: Quadriceps Exercise Before Total Knee Arthroplasty (The QUADX-1 Trial)
Acronym: QUADX-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Rasmus Skov Husted, PhD, MSc., PT., Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HvidovreUH - QUADX-1 Trial
Record Dates: First submitted 2016-10-03; First posted 2016-10-12 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee-extension exercise; Quadriceps exercise; Knee osteoarthritis; Exercise adherence; Dose-response relationship; Prehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 2 (Active Comparator): Two knee-extension exercise sessions per week. Each exercise session comprises a single strength training exercise; knee-extension, which is performed in 3 sets with 12 RM repetitions in each set.
  The knee-extension resistance training exercise is performed with an elastic exercise band.
  Interventions: Other: Two knee-extension exercise sessions per week.
- Group 4 (Active Comparator): Four knee-extension exercise sessions per week. Each exercise session comprises a single strength training exercise; knee-extension, which is performed in 3 sets with 12 RM repetitions in each set.
  The knee-extension resistance training exercise is performed with an elastic exercise band.
  Interventions: Other: Four knee-extension exercise sessions per week.
- Group 6 (Active Comparator): Six knee-extension exercise sessions per week. Each exercise session comprises a single strength training exercise; knee-extension, which is performed in 3 sets with 12 RM repetitions in each set.
  The knee-extension resistance training exercise is performed with an elastic exercise band.
  Interventions: Other: Six knee-extension exercise sessions per week.

INTERVENTIONS:
Other: Two knee-extension exercise sessions per week. — Each exercise session comprises a single strength training exercise; knee-extension, which is performed in 3 sets with 12 RM repetitions in each set.
  The knee-extension resistance training exercise is performed with an elastic exercise band.
  Arms: Group 2
Other: Four knee-extension exercise sessions per week. — Each exercise session comprises a single strength training exercise; knee-extension, which is performed in 3 sets with 12 RM repetitions in each set.
  The knee-extension resistance training exercise is performed with an elastic exercise band.
  Arms: Group 4
Other: Six knee-extension exercise sessions per week. — Each exercise session comprises a single strength training exercise; knee-extension, which is performed in 3 sets with 12 RM repetitions in each set.
  The knee-extension resistance training exercise is performed with an elastic exercise band.
  Arms: Group 6

SUMMARY:
The trial investigates the efficacy of knee-extension exercise prior to total knee replacement. The participants are randomly allocated to one of three exercise dosages. There is no control group.

DETAILED DESCRIPTION:
Patients with end-stage knee osteoarthritis (OA) have decreased knee-extension strength and suffer from knee pain. Strengthening of the knee-extensor muscle is a key element in conservative treatment for patients with knee OA. However, the most effective exercise dosage for knee-extension strength exercise is unknown.

In this trial the investigators investigate the efficacy of three different dosages of knee-extension strength exercise. Patients eligible for total knee replacement are offered home-based pre-operative knee-extension exercise and are randomly allocated to one of three exercise dosage groups. There is no control group. The knee-extension exercise is performed with an elastic exercise band mounted with sensor (BandCizer) which registers when the patients exercise, how much they exercise and how they exercise.

The intervention time is 12 weeks and the primary time point of interest is after exercise/just before surgery. Secondary time points of interest are shortly after surgery and three months after surgery.

The patients are given detailed exercise instruction at trial entry and hereafter they exercise unsupervised at home for 12 weeks. At week 4 and 8 they receive follow-up instruction.

Both the patients who choose not to have TKA and those who do after the exercise period will be followed with annual outcome assessments as part of a follow-up cohort.

Embedded in the trial is a qualitative study. Focus group interviews will be performed with the participating patients about their experienced enablers and barriers related to adherence to the home-based intervention, once the post-operative outcome assessment has been completed. Likewise, the orthopedic surgeons and physiotherapists allocated to the trial will undergo focus group interviews, once the trial is completed, to explore their experienced enablers and barriers related to administering the home-based intervention.

Protocol amendments 8/2-2017: Additional protocol approved by The Danish National Committee on Biomedical Research Ethics (protocol no. 55528 and 55529). Approved protocol amendments are the following inclusion and exclusion criteria: inclusion criteria age ≥45, and exclusion criteria ASA-score ≥4.

Protocol amendments 30/3-2017: Additional protocol approved by The Danish National Committee on Biomedical Research Ethics (protocol no. 57312). Approved protocol amendments are the following inclusion criteria: knee pain during the last week (NRS) ≥3, and the OKS questionnaire score has been omitted as an inclusion criteria.

Protocol amendments 6/9-2017: At the third outcome assessment (at hospital discharge, 3-8 days after surgery) only the outcomes isometric knee-extensor strength, 6MWT, SCT and current knee pain are assessed. The KOOS and OKS questionnaires as well as knee pain during the last week are omitted at this end-point as they are not validated to assess acute post-operative conditions, and use a too long recall period.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a possible candidate for a primary TKA due to knee osteoarthritis
* Patient is eligible for home-based quadriceps exercise
* Patient has an age ≥ 50 years
* Patient is a possible candidate for primary unilateral TKA, based on all the below terms:

  * Knee pain >3 (Numeric Rating Scale) in the last week
  * Kellgren-Lawrence classification grade ≥2
  * Oxford Knee Score <30
* Patient is resident in one of the three municipalities (København, Hvidovre or Brøndby) involved in the trial
* Patient is able to speak and understand Danish

Exclusion Criteria:

* Exercise is contra-indicated for the patient
* Patient has a neurological disorder
* Patient has a diagnosed systemic disease (ASA score ≥ 3)
* Patients with terminal illness
* Patient has severe bone deformity demanding use of nonstandard implants
* Weekly alcohol consumption above national recommendations (>7 units women, >14 units men)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Isometric knee-extension strength at 60 degrees knee flexion measured as Nm/kg body mass | Change from 1) baseline to 2) after 12 weeks of exercise/just before surgery
  The measurement will be assessed using a computerized strength chair (Good Strength Chair, Metitur Oy, Jyvaskyla, Finland).

SECONDARY OUTCOMES:
Isometric knee-extension strength at 60 degrees knee flexion measured as Nm/kg body mass | Change from 1) baseline to 3) at hospital discharge (3-8 days after surgery), and change from 1) baseline to 4) three months after surgery
  The measurement will be assessed using a computerized strength chair (Good Strength Chair, Metitur Oy, Jyvaskyla, Finland).
6 min walk test for distance (6MWT) | Change from 1) baseline to 2) after 12 weeks of exercise/just before surgery, and change from 1) baseline to 3) at hospital discharge (3-8 days after surgery), and change from 1) baseline to 4) three months after surgery
  The test measures the maximal distance a participant is able to walk in six minutes between two cones placed 29 meters apart from each other.
Stair climb test (SCT) | Change from 1) baseline to 2) after 12 weeks of exercise/just before surgery, and change from 1) baseline to 3) at hospital discharge (3-8 days after surgery), and change from 1) baseline to 4) three months after surgery
  The test measure the time (seconds) it takes to ascend and descend an 11-step flight of stairs with 16 cm step height.
Knee Osteoarthritis Outcome Score (KOOS) | Change from 1) baseline to 2) after 12 weeks of exercise/just before surgery, and change from 1) baseline to 3) at hospital discharge (3-8 days after surgery), and change from 1) baseline to 4) three months after surgery
  The KOOS is a questionnaire with 42 questions regarding knee function.
Oxford Knee Score (OKS) | Change from 1) baseline to 2) after 12 weeks of exercise/just before surgery, and change from 1) baseline to 3) at hospital discharge (3-8 days after surgery), and change from 1) baseline to 4) three months after surgery
  The OKS is a 12-item questionnaire regarding knee related function and pain in patients with knee OA.
Knee pain | Change from 1) baseline to 2) after 12 weeks of exercise/just before surgery, and change from 1) baseline to 3) at hospital discharge (3-8 days after surgery), and change from 1) baseline to 4) three months after surgery
  Individual knee pain is assessed with the Numeric Rating Scale (NRS). This is an 11-point subjective pain scale ranging from 0-10 (0 indicating no pain).
Surgical status | Assessment at 2) after 12 weeks of exercise/just before surgery
  At the 2nd outcome assessment (after the 12 weeks exercise period) the patients are asked by the outcome assessor "based on your knee symptoms in the last week would you say that you need knee surgery now?" The answer will be categorized into one of three options; 1) 'yes' I believe I need surgery now, 2) I do not know or, 3) 'no' I do not believe I need surgery now.
Exercise adherence | Assessment at 2) after 12 weeks of exercise/just before surgery
  Adherence to the home-based single knee-extension strength exercise will be assessed with elastics exercise bands with build-in BandCizer (sensor) technology.The sensor stores data on date, time, number of sets, repetitions, tonnage (kg x repetitions), and time-under-tension (TUT). In the present trial, a patient is defined as adherent to the exercise intervention if >75% of the prescribed exercise sessions are completed.

OTHER OUTCOMES:
Adverse events | Assessment at 2) after 12 weeks of exercise/just before surgery, 3) at hospital discharge (3-8 days after surgery) and 4) three months after surgery
  All adverse events occurring while the patient is enrolled in the trial will be recorded regardless of its relation to the exercise intervention, surgery or occurrences not related to the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bandholm, PhD, Study Director — Clinical Research Center, Hvidovre University Hospital; Rasmus S Husted, MSc., PT., Principal Investigator — Clinical Research Center, Hvidovre University Hospital
Locations (1):
- Clinical Research Centre, Amager Hvidovre hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Husted RS, Troelsen A, Husted H, Gronfeldt BM, Thorborg K, Kallemose T, Rathleff MS, Bandholm T. Knee-extensor strength, symptoms, and need for surgery after two, four, or six exercise sessions/week using a home-based one-exercise program: a randomized dose-response trial of knee-extensor resistance exercise in patients eligible for knee replacement (the QUADX-1 trial). Osteoarthritis Cartilage. 2022 Jul;30(7):973-986. doi: 10.1016/j.joca.2022.04.001. Epub 2022 Apr 9. PMID 35413476
- [Derived] Husted RS, Bandholm T, Rathleff MS, Troelsen A, Kirk J. Perceived facilitators and barriers among physical therapists and orthopedic surgeons to pre-operative home-based exercise with one exercise-only in patients eligible for knee replacement: A qualitative interview study nested in the QUADX-1 trial. PLoS One. 2020 Oct 23;15(10):e0241175. doi: 10.1371/journal.pone.0241175. eCollection 2020. PMID 33095777
- [Derived] Husted RS, Troelsen A, Thorborg K, Rathleff MS, Husted H, Bandholm T. Efficacy of pre-operative quadriceps strength training on knee-extensor strength before and shortly following total knee arthroplasty: protocol for a randomized, dose-response trial (The QUADX-1 trial). Trials. 2018 Jan 18;19(1):47. doi: 10.1186/s13063-017-2366-9. PMID 29347947
- See also: Physical Medicine & Rehabilitation Research - Copenhagen (PMR-C) — https://www.hvidovrehospital.dk/pmr-c/Pages/default.aspx?rhKeywords=pmr
- Available data/document: Study Protocol — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-017-2366-9
- Available data/document: Clinical Study Report — https://www.clinicalkey.com/#!/content/journal/1-s2.0-S1063458422007154